CLINICAL TRIAL: NCT07041346
Title: The Effect of Gender Education Provided to Health Sciences Students on Gender Perception and Roles: A Randomized Controlled Trial
Brief Title: The Effect of Gender Education Provided to Health Sciences Students on Gender Perception and Roles
Acronym: Education
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Beyzanur İşbay Aydemir, Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/07
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: EDUCATION
Keywords: Gender education; Gender perception; Gender roles
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: Education
- No Intervention (No Intervention)

INTERVENTIONS:
Other: Education — 1. Objectives of the Training Program To increase students' knowledge and awareness of gender concepts, gender roles, and gender inequality.
     To help students develop more conscious and critical thinking skills regarding social norms and gender-based discrimination.
     To promote the development of gender-sensitive attitudes and contribute to positive attitude changes following the training.
  2. Duration and Structure of the Training Total Duration: 2 weeks
     Weekly Duration: 2 hours
     Training Format: In-person
     Training Methods: Presentations, group discussions, surveys, brainstorming, Q&A sessions, debates
  3. Training Content and Modules Week 1 Topic 1: Fundamental Concepts, Gender Roles, and Inequality
  Introduction and Training Objectives
  Gender and Social Norms: Definition of gender norms and their impact on individuals
  Arms: Experimental

SUMMARY:
Sexual health is a fundamental component of living a healthy and fulfilling life. However, in societies where sexual health education is inadequate, factors such as social norms and gender inequality hinder individuals from properly understanding sexual health and developing healthy sexual behaviors. The gender roles established by society and the stereotypes associated with these roles shape individuals' sexual identities and experiences, often based on narrow and rigid views of masculinity and femininity. In societies where gender roles are strictly defined, such norms can place serious limitations on individuals' sexual rights, freedoms, and ability to form healthy relationships.

In this context, sexual health education plays a vital role in raising awareness about societal norms and helping transform these norms. Gender inequality is another major barrier that complicates the accurate understanding of sexual health. In many communities, especially for women, sexual rights are limited due to cultural values, traditional beliefs, and social pressures. This restricts their access to sexual health services and their ability to protect themselves.

Sexual health education aims to eliminate these inequalities and ensure that all individuals, regardless of gender, can maintain a healthy sexual life with equal rights. These educational efforts not only create awareness about gender inequality but also support the promotion of healthy and safe sexual behaviors.

DETAILED DESCRIPTION:
Implementation of the Study

Participants will be informed that no financial compensation will be provided for participation, and this will be clearly stated in the written informed consent form.

Following the approval of the ethics committee, institutional permission will be obtained from Istanbul Aydın University, where the study will be conducted. The study will take place at the Faculty of Health Sciences, where one of the researchers, Beyzanur İşbay Aydemir, is affiliated.

Students enrolled in various departments (e.g., Nursing, Physiotherapy and Rehabilitation, Audiology) within the Faculty of Health Sciences who voluntarily agree to participate will be included in the study.

Data will be collected using a Diagnostic Form, the Gender Perception Scale, and the Attitude Scale Towards Gender Roles. Participants who agree to join the study will be fully informed by the researcher about the purpose, scope, and procedures of the research. After this briefing, both verbal and written informed consent will be obtained, and the forms will be completed.

To inform and invite students to the study, a research announcement poster will be prepared and displayed on bulletin boards throughout the Faculty of Health Sciences campus.

In addition, faculty members teaching in relevant departments will be asked to provide a brief explanation of the study during class and to encourage student participation. This strategy aims to increase awareness of the study and reach a broader group of students.

The research will utilize a pre-test-post-test control group experimental design. Students who provide informed consent and meet the inclusion criteria will be randomly assigned to the experimental and control groups using the simple randomization method.

This random assignment will be conducted using computer-based software (e.g., randomizer.org), ensuring an unbiased and balanced distribution across the study groups.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in a department within the Faculty of Health Sciences

Being 18 years of age or older

Voluntarily agreeing to participate in the study

Exclusion Criteria:

* Failing to complete the study after initially agreeing to participate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Gender Perception Scale | 5 minutes
  The Gender Perception Scale (GPS) is a 25-item, 5-point Likert-type scale (1 = strongly disagree, 5 = strongly agree) developed to assess individuals' perceptions of gender. The scale includes both positively worded items (10 items), such as "Marriage does not prevent a woman from working" and "Working women can also spend enough time with their children", as well as negatively worded (reverse scored) items (15 items), such as "A woman should not work if her husband does not allow it" and "A woman without a husband is like a house without an owner."
  The total score ranges from 25 to 125. Higher scores indicate a more egalitarian perception of gender roles. Exploratory factor analysis revealed that the scale has a unidimensional structure. The internal consistency reliability of the scale, as measured by Cronbach's alpha, is .87.
Attitude Scale Toward Gender Roles | 5 minutes
  The Attitude Scale Toward Gender Roles was originally developed by García-Cueto et al. in 2015 and was adapted into Turkish by Bakioğlu and Türküm in 2019. The scale aims to assess individuals' egalitarian attitudes toward gender roles. It consists of 15 items and is structured as a unidimensional, 5-point Likert-type scale (1 = strongly disagree; 5 = strongly agree).
  The last 13 items of the scale are reverse-coded, and the total score is calculated by summing all item scores after the necessary recoding. Higher total scores indicate a more egalitarian attitude toward gender roles.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Şahin Tokatlıoğlu, PhD, Study Chair — bisbay1694@gmail.com; Nur Bahar KURU AKTURK, Msc, Study Chair — nurbaharkuru@arel.edu.tr; Gül DİKEÇ, Assoc. Prof., Study Chair — guloban@hotmail.com
Locations (1):
- Sağlık Bilimleri Ünversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No